CLINICAL TRIAL: NCT03558763
Title: Remote MONITORing of Patients With Chronic Obstructive Pulmonary Disease Using a Tablet System. A Randomized Cross Over Pilot Study of Feasibility Evaluation and Quality of Life Measurements
Brief Title: Remote Monitoring of Patients With COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MONITOR
Record Dates: First submitted 2018-05-23; First posted 2018-06-15 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-05

CONDITIONS: COPD
Keywords: Monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This clinical trial is an open, randomized, controlled cross-over study. Eligible subjects to include will be given the possibility to participate in the study. They will at their first visit be randomized to start either telemonitoring, using the tablet system arm or to normal standard of care period for 26 weeks. After 26 weeks the subject will have a second visit and after that, four weeks (wash out) of standard of care or telemonitoring treatment. After that there will be a third visit and the subject will start the second treatment period with the alternative management. At the end of this period (56 weeks) there will be a fourth (last) visit at the center for the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Care (Active Comparator): During normal care the subjects will get the possibility to call the COPD-center via telephone on their own initiative e g with worsening symptoms as usual.
  Interventions: Other: Normal Care
- Telemonitoring (Active Comparator): Twice a week subject will perform additional vital functions:
  Blood pressure and heart rate will be measured using the Electronic Sphygmomanometers "Track".
  Weight will be taken using the Scale "lite" Oxygen saturation will be measured using Pulse Oximeter "Air" And
  Complete two PRO´s (integrated in the application):
  CAT MRC All this is estimated to take approximately 20-30 min each time.
  For the first 4 weeks there will be weekly video calls with a COPD-center nurse discussing health condition and vital parameters.
  Thereafter there will be monthly video calls with a COPD-center nurse for the remaining 5 months, i.e. 4 further calls. The video calls will take approximately 15 min.
  Interventions: Device: Telemonitoring

INTERVENTIONS:
Device: Telemonitoring — During the telemonitoring treatment period the subjects will register; vital functions (blood pressure, heart rate, weight, SpO2) twice a week, physical movement daily by using a fitness device, have video calls with a nurse weekly the first 4 weeks and thereafter every fourth week the last 5 months. Twice a week (± 2 days) questionnaires (CAT and MRC) should be filled out at home.
  Arms: Telemonitoring
Other: Normal Care — During normal care the subjects will get the possibility to call the COPD-center via telephone on their own initiative e g with worsening symptoms as usual.
  Arms: Normal Care

SUMMARY:
This clinical investigation will evaluate the patient-equipment interface and patient preference in the use of modern possibilities for remote monitoring of patients with COPD in a personalized care approach.

DETAILED DESCRIPTION:
The primary objective is to evaluate the impact and feasibility of tele monitoring and video contact in personalized care of moderate and severe COPD patients. This should be compared to normal standards of care. The cross-over design evaluates the influence on general HRQOL of this tablet and monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and provision of informed consent
* Diagnosis of COPD
* FEV1/FVC (post bronchodilator) <0.7
* GOLD severity grade D
* FEV, < 80% predicted
* Cognitive ability relevant for the studies as judged by the investigator
* Living in their own home and able to manage their activities of daily living

Exclusion Criteria:

* Rapidly progressing severe disease other than COPD and COPD-related diseases, influencing the Health-Related Quality of Life (HRQOL) during the study time as judged by the investigator
* Long-term stay ( >2 weeks) away from home during the study period, where there are no possibility to get internet connection
* COPD exacerbation during 1 month before start of study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change of SF-12 over each treatment period | 13 month study, measure points at day 0 (1), week 26 (2), week 30 (3) and week 56 (4)
  The primary objective is to evaluate the impact and feasibility of tele monitoring and video contact in personalized care of moderate and severe COPD patients. This should be compared to normal standards of care. The cross-over design evaluates the influence on general HRQOL of this tablet and monitoring system.

OTHER OUTCOMES:
Cost-utility evaluation | 13 months
  The difference in costs between the two treatments divided by the difference in quality adjusted life years (QALYs)
  For other secondary measures: Descriptive statistics will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Ullman, MD Phd, Principal Investigator — Head of COPD center; Lowie Vanfleteren, MD Phd, Principal Investigator — Head of COPD center
Locations (1):
- COPD center, Gothenburg, Västra Götaland County, Sweden

DOCUMENTS (1):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03558763/Prot_000.pdf